CLINICAL TRIAL: NCT07045311
Title: JS207 Combination Therapy in Recurrent or Metastatic Triple-negative Breast Cancer(TNBC)
Brief Title: JS207 Combination Therapy in Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS207-008-II-TNBC
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Masking Description: None(open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental)
  Interventions: Drug: JS207 in combination with 9MW2821
- Cohort B (Experimental)
  Interventions: Drug: JS207 in combination with Albumin paclitaxel

INTERVENTIONS:
Drug: JS207 in combination with 9MW2821 — JS207 will be administered intravenously at a dose of 10 mg/kg (D1, Q3W), 9MW2821 will be administered intravenously at a dose of 1.25 m.g/kg (D1 and D8, Q3W)
  Arms: Cohort A
Drug: JS207 in combination with Albumin paclitaxel — JS207 will be administered intravenously at a dose of 10 mg/kg (D1, Q3W), Albumin paclitaxel will be administered intravenously at a dose of 125 mg/m2 (D1 and D8, Q3W).
  Arms: Cohort B

SUMMARY:
This is an open-label, multi-center, phase II clinical study to preliminarily evaluate the efficacy and safety of JS207 combined with 9MW2821 or albumin paclitaxel as first-line therapy in patients with recurrent or metastatic TNBC.

DETAILED DESCRIPTION:
The study consists of Cohort A and Cohort B. Both cohorts include patients with recurrent or metastatic TNBC who have not received systemic anti-tumor therapy previously. Cohort A will receive JS207 combined with 9MW2821, and Cohort B will receive JS207 combined with albumin paclitaxel. Each cohort consists of two stages: safety run-in period and cohort expansion period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 - 75 years old；
2. Voluntary participation in clinical study；
3. Histologically confirmed unresectable, locally advanced or metastatic triple-negative breast cancer(absence of HER2, ER, and PR expression);
4. No prior systemic antitumor therapy for locally advanced or Metastatic TNBC；
5. Prior use of systemic anti-tumor therapy in the neoadjuvant and/or adjuvant phase is allowed, but must meet the following conditions: (1) the time interval between the end of neoadjuvant/adjuvant therapy and the occurrence of recurrence/metastasis is ≥6 months; (2) Arm2: if taxane is used in the neoadjuvant/adjuvant phase, the DFI must be ≥12 months;
6. Adequate organ function;
7. ECOG performance status of 0 or 1;
8. Life expectancy 12 weeks;
9. Measurable disease, as defined by RECIST v1.1;

Exclusion Criteria:

1. Untreated or active central nervous system (CNS) metastases；
2. Uncontrolled pleural effusion, pericardial effusion or ascites；
3. Tumor encasement of important vessels or significant necrosis and cavitation that may cause a risk of hemorrhage；
4. History of significant bleeding tendency or severe coagulation disorder；
5. Uncontrolled hypertension；
6. Active autoimmune diseases requiring systemic treatmen within 2 years prior to the first dose；
7. History of interstitial lung disease or previous Noninfectious pneumonitis treated with corticosteroids, or evidence of active Pneumonia in radiology on screening period；
8. Eye disorders or symptoms: severe xerophthalmia, keratoconjunctivitis sicca, severe exposure keratitis, or other conditions；
9. Severe cardiovascular disease；
10. Serious infection (CTCAE 5.0 Grade>2) within 28 days prior to the first dose of study drug；
11. Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs targeting other stimulatory or co-inhibitory T cell receptors (e.g., CTLA-4, OX-40, CD137) in (new) adjuvant therapy is allowed, if DFI is ≥6 months previously treated with Antibody-Drug Conjugates conjugated with MMAE and/or targeting Nectin-4, such as Enfortumab Vedotin is not allowed；
12. History of another malignancy within 5 years before the first dose of study drug；
13. Not suitable to receive study treatment for other conditions as per investigator；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-03-22 (Estimated); Study Completion 2029-03-22 (Estimated)

PRIMARY OUTCOMES:
ORR | 2years
  Objective response rate（ORR） evaluated based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria

SECONDARY OUTCOMES:
DOR | 2years
  Duration of response (DoR) evaluated based on RECIST v1.1
DCR | 2years
  Disease control rate (DCR) evaluated based on RECIST v1.1
PFS | 2years
  Progression-free survival (PFS) evaluated based on RECIST v1.1
OS | 3years
  The time from first dose to death from any cause
AE | 2years
  Incidence and severity of Adverse Events(AEs)according to NCI-CTCAE v5.0
Plasma concentrations | 2years
  Plasma concentrations of JS207 and 9MW2821.
ADA | 2years
  The incidence and titer of anti-drug antibodies (ADA) of JS207 and 9MW2821
Nab | 2years
  The incidence of Nab(if applicable) of JS207 and 9MW2821
PD-L1 | 2years
  The correlation between PD-L1 expression in tumor tissue and therapeutic efficacy
Nectin-4 | 2years
  The correlation between Nectin-4 expression in tumor tissue and therapeutic efficacy

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Guangdong women and children's hospital and health institute, Guangzhou, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Affiliated Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhangzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanchang People'S Hospital, Nanchang, Jiangxi
  - Jilin University First Hospital, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - Ceneral Hosipital of Ningxia Medical University, Yinchuan, Ningxia
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Xi'an International Medical Center Hospital, Xian, Shanxi
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No